CLINICAL TRIAL: NCT01102946
Title: Panretinal Photocoagulation Versus Panretinal Photocoagulation Plus Intravitreous Ranibizumab for High Risk Proliferative Diabetic Retinopathy
Brief Title: Panretinal Photocoagulation (PRP) Plus Ranibizumab for Proliferative Diabetic Retinopathy
Acronym: IRaHi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Rodrigo Jorge, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRaHi
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-01

CONDITIONS: Diabetic Retinopathy; Retinal Neovascularization
Keywords: proliferative diabetic retinopathy; retinal neovascularization; Angiogenesis Inhibitors; ranibizumab; laser
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRP plus ranibizumab (Experimental): Patients will be submitted to panretinal photocoagulation plus intravitreal injections of ranibizumab
  Interventions: Drug: Ranibizumab; Procedure: Panretinal Photocoagulation
- PRP (Active Comparator): Patients will only be submitted to panretinal photocoagulation
  Interventions: Procedure: Panretinal Photocoagulation

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab (Lucentis), intravitreal injections of 0.05ml
  Other Names: Lucentis
  Arms: PRP plus ranibizumab
Procedure: Panretinal Photocoagulation — Panretinal photocoagulation with green laser according to ETDRS

SUMMARY:
The purpose of this study is to evaluate the effects of panretinal photocoagulation plus intravitreal ranibizumab for the treatment of patients with high risk proliferative diabetic retinopathy in terms of changes in visual acuity and neovascularization area.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* High risk proliferative diabetic retinopathy
* Visual acuity ≥ 20/800
* No previous laser treatment for diabetic retinopathy

Exclusion Criteria:

* Previous pars plana vitrectomy
* Systemic thrombo-embolic events
* Uncontrolled systemic hypertension
* Conditions avoiding adequated documentation
* Previous eye surgery in the last 6 months before inclusion in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Fluorescein leakage area (mm2) | Week 48 after inclusion in the study
  Neovascularization area measured during fluorescein agiography middle phase

SECONDARY OUTCOMES:
CMT | Week 48 after inclusion in the study
  Macular thickness measured with Stratus OCT protocols
LogMAR BCVA | Week 48 after inclusion in the study
  LogMAR best corrected visual acuity measured with ETDRS charts
Retina mid periphery visual field sensitivity change | Week 48 after inclusion in the study
Rod pathway integrity and oscillatory potential amplitudes | Week 48 after inclusion in the study

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: article on Pubmed — http://www.ncbi.nlm.nih.gov/pubmed/21726427